CLINICAL TRIAL: NCT05768464
Title: A Prospective, Multicenter, Single-arm Clinical Study of the Efficacy and Safety of Toripalimab in Combination With Axitinib for Postoperative Adjuvant Therapy for Non-clear Renal Cell Carcinoma With High-risk Recurrence Factors
Brief Title: Postoperative Adjuvant Therapy for Non-clear Renal Cell Carcinoma With High-risk Recurrence Factors
Acronym: IUNU-RC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-RC-102
Record Dates: First submitted 2022-12-17; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-12

CONDITIONS: Non-clear Renal Cell Carcinoma
Keywords: toripalimab; axitinib; postoperative adjuvant therapy
MeSH Terms: interventions — toripalimab; spartalizumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Drug: Toripalimab 240mg, intravenously every 3 weeks
  Drug: Axitinib 5 mg orraly twice daily
  Interventions: Drug: Toripalimab; Drug: Axitinib

INTERVENTIONS:
Drug: Toripalimab — 240mg intravenously every 3 weeks
  Other Names: anti-PD-1 monoclonal antibody
Drug: Axitinib — 5mg orraly twice daily
  Other Names: TKI

SUMMARY:
The goal of this prospective, multicenter, single-arm clinical study is to evaluate the efficacy and safety of toripalimab in combination with axitinib for postoperative adjuvant therapy for non-clear renal cell carcinoma with high-risk recurrence factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Participants with histologically confirmed non-clear renal cell carcinoma except clear cell RCC, chromophobe RCC and eosinophilic RCC, and must meet any of the following conditions:

   1. histologically confirmed Papillary RCC, pT≥T1b and ISUP/WHO ≥3, N (any), M0;
   2. Collecting duct carcinoma, SMARCB1-deficient renal medullary carcinoma, fumarate hydratase deficiency renal cell carcinoma (FH-RCC), pT (any), ISUP/WHO (any), N (any), M0.
   3. Non-clear renal cell carcinoma except Organizational Credits Type a and b, including but not limited to TFE3/TFEB translocated RCC or unclassified RCC, pT (any), ISUP/WHO ≥ grade 3, N (any), M0;
3. Patients who have completely resected the primary tumor (partial or radical nephrectomy), and M1 NED patients who have completely resected solid, isolated soft tissue metastases.
4. Patients who have completely removed the renal tumor. The nephrectomy must be performed ≥ 3 weeks but ≤ 12 weeks before randomization. Partial nephrectomy and renal tumor enucleation are permitted;
5. Patients must have no clinical or radiographic evidence of macroscopic residual lesions or distant metastasis (M0) after surgery. M1 participants must have no evidence of disease (M1 NED);
6. ECOG performance status 0-1 ;
7. Patients must have not received systemic therapy for renal tumors;
8. Adequate hematopoiesis and organ function:

   * Hematopoietic function: Absolute neutrophil count (ANC) ≥1.5×109/L; platelets≥ 100×109/L; Hemoglobin≥ 9.0g/dL;
   * Renal function: serum creatinine ≤ 1.5 times ULN, or creatinine clearance > 50 mL/min;
   * Liver function: total bilirubin ≤1.5×ULN or total bilirubin >1.5×ULN but direct bilirubin normal; AST and ALT≤2.5×ULN;
   * Coagulation function: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN;
   * Left ventricular ejection fraction (LVEF) ≥ 50%;
9. Signed informed consent form;
10. Patients and/or their partner are willing to use highly effective forms of contraception and to continue its use 3 months after the last dose of drugs.
11. Ability and capacity to comply with study and follow-up procedures.

Exclusion Criteria:

1. Clear cell RCC, chromophobe RCC and eosinophilic RCC;
2. Previous anti-tumor immunotherapy, including but not limited to cytokines (IL-2, IFN-α, etc.) and antibody drugs (anti-PD-1, PD-L1, or CTLA-4 antibodies, etc.)
3. Previous drug therapy targeting VEGF, VEGFR, or mTOR;
4. Have participated in or are currently participating in an investigational drug trial within 4 weeks; major surgery performed within 4 weeks prior to randomization;
5. Receive traditional Chinese medicines or proprietary Chinese medicine, adrenocortical hormone or other immunosuppressant systemic therapy within 2 weeks before enrollment; People who > 10 mg of prednisone or equivalent inhalers daily but have no active autoimmune disease may participate in this study;
6. Toxicity has not been relieved after previous antineoplastic therapy; Irreversible toxicities (e.g., hearing loss) that are reasonably expected not to be aggravated by the study drug may participate in this study;
7. Other malignancies that have progressed or require treatment in 5 years (excluding adequately treated basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, superficial bladder cancer, breast, cervix, or prostate carcinoma in situ);
8. History of central nervous system (CNS) metastases or CNS metastases on baseline imaging (MRI or CT) within 30 days prior to the first trial administration;
9. Hypertension that cannot be controlled by medications (blood pressure 150/100 mmHg despite optimal medical therapy)
10. Evidence of following cardiovascular disease within 6 months:

    1. Myocardial infarction
    2. Unstable angina
    3. Cardiac angioplasty or stenting
    4. Coronary/peripheral artery bypass grafting
    5. Class III or IV congestive heart failure as prescribed by the New York Heart Association
    6. Cerebrovascular accident or transient ischemic attack
11. QT interval (QTc) corrected with heart rate ≥500 msec (Bazett's formula)
12. History of active or other severe bleeding within 30 days, and have haemoptysis within 6 weeks prior to randomization;
13. Deep vein thrombosis or pulmonary embolism within 6 months;
14. Clinically significant gastrointestinal (GI) abnormalities, including:

    1. malabsorption, total gastrectomy or any condition that may affect the absorption of oral medications;
    2. active ulcers treated within the past 6 months;
    3. active gastrointestinal bleeding (e.g., hematemesis, hematochezia, or melena) within the past 3 months with no evidence of healing endoscopic or colonoscopy;
    4. Metastatic lesions of the gastrointestinal tract suspected of bleeding, inflammatory bowel disease, ulcerative colitis, perforation of the digestive tract or other gastrointestinal diseases that increase the risk of perforation;
15. History of organ transplantation may require long-term adrenocortical hormone therapy;
16. Previous or current presence of (noninfectious) pneumonia/interstitial lung disease requiring adrenocortical hormone therapy
17. Active infection requiring systemic treatment, human immunodeficiency virus (HIV) infection (known HIV antibody positive), active HBV or HCV infection;
18. Have received a live vaccine within 30 days prior to enrollment;
19. History of severe drug allergy;
20. Known history of psychiatric illness or substance abuse;
21. The presence of unhealed wounds;
22. Taken within 7 days prior to enrollment or expected to take concomitant treatment with potent CYP3A4/5 inhibitors and CYP3A4/5 inducers ;
23. Subject has a history or current evidence of any disease, treatment, or laboratory abnormality that may confound the trial results, interfere with the subject's participation in the full trial, or is not in the best interest of the subject to participate in the trial, in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
DFS | 2 years
  DFS is defined as time interval from the date of randomization to first date of recurrence/relapse (distant or local recurrence of [RCC] or occurrence of a secondary malignancy {occurrence of a second primary cancer other than RCC} or death). For participants with no DFS event, DFS was censored at date of last scan prior to time of analyses. Participants alive who did not have post-baseline disease assessments, DFS was censored at randomization. Participants who received further anti-tumor therapy prior to recurrence or occurrence of a secondary malignancy or death, DFS was censored on date of last scan prior to taking anti-tumor medication. Participants who missed 2 or more consecutive tumor scans immediately followed by an event were censored at date of last objective tumor assessment prior to missing/not readable scan.

SECONDARY OUTCOMES:
OS | 3 years
  OS defined as the time from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. Participants lacking data beyond randomization had their survival times censored at randomization.
DRSS | 3 years
  Localised disease recurrence-specific survival
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Incidence and grade of AEs and SAEs per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, incidence of ≥ grade 3 AE

CONTACTS AND LOCATIONS:
Overall Officials: hongqian guo, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (2):
- China (2):
  - Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu
  - Hongqian Guo, Nanning, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu T, Zhang M, Sun D. Immune Cell Infiltration and Identifying Genes of Prognostic Value in the Papillary Renal Cell Carcinoma Microenvironment by Bioinformatics Analysis. Biomed Res Int. 2020 Jul 25;2020:5019746. doi: 10.1155/2020/5019746. eCollection 2020. PMID 32775427
- [Background] Lobo J, Ohashi R, Amin MB, Berney DM, Comperat EM, Cree IA, Gill AJ, Hartmann A, Menon S, Netto GJ, Raspollini MR, Rubin MA, Tan PH, Tickoo SK, Tsuzuki T, Turajlic S, Zhou M, Srigley JR, Moch H. WHO 2022 landscape of papillary and chromophobe renal cell carcinoma. Histopathology. 2022 Oct;81(4):426-438. doi: 10.1111/his.14700. Epub 2022 Jun 10. PMID 35596618
- [Background] Steffens S, Janssen M, Roos FC, Becker F, Schumacher S, Seidel C, Wegener G, Thuroff JW, Hofmann R, Stockle M, Siemer S, Schrader M, Hartmann A, Kuczyk MA, Junker K, Schrader AJ. Incidence and long-term prognosis of papillary compared to clear cell renal cell carcinoma--a multicentre study. Eur J Cancer. 2012 Oct;48(15):2347-52. doi: 10.1016/j.ejca.2012.05.002. Epub 2012 Jun 13. PMID 22698386